CLINICAL TRIAL: NCT00225732
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial of Ibuprofen Injection (IVIb) for Treatment of Pain in the Post-Operative Adult Patients
Brief Title: Trial of Caldolor for Treatment of Pain in Post-Operative Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPI-CL-008
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Results first posted 2011-09-15 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous ibuprofen (Active Comparator)
  Interventions: Drug: Intravenous ibuprofen
- normal saline (Placebo Comparator)
  Interventions: Other: Normal saline as placebo comparator

INTERVENTIONS:
Other: Normal saline as placebo comparator — 250 ml normal saline as a placebo comparator was administered every 6 hours for a total of eight doses over the first 48 hours. Those patients who received the initial eight doses could continue to receive additional doses as needed through the end of the treatment period (day 5)
  Other Names: NS
  Arms: normal saline
Drug: Intravenous ibuprofen — 800 mg intravenous ibuprofen diluted in 250 milliliters of normal saline was administered every 6 hours for a total of eight doses over the first 48 hours.
  Those patients who received the initial eight doses could continue to receive additional doses as needed through the end of the treatment period (day 5)
  Other Names: Caldolor
  Arms: intravenous ibuprofen

SUMMARY:
The primary objective of this study of Caldolor (IV ibuprofen) administered to post-operative hospitalized adult patients every 6 hours for 48 hours is to determine the efficacy of Caldolor compared to placebo for the treatment of post-operative pain as measured by reduction in the requirement for the narcotic analgesic, morphine, post surgery

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for elective abdominal hysterectomy surgery with anticipated need for post-operative I.V. morphine analgesia with anticipated use of ≥ 24 hours.
2. Adequate IV access
3. Anticipated hospital stay ≥ 24 hours

Exclusion Criteria:

1. Be unable to make a reliable self-report of pain intensity to pain relief
2. Less than 18 years of age
3. Greater than 70 years of age
4. Use of NSAIDs within 12 hours prior to dosing
5. Use of analgesics, muscle relaxants and sedatives less than 24 hours prior to CTM administration with the following exceptions: paracetamol (acetaminophen) can be administered until 6 hours prior to surgery; tramadol can be administered until midnight the evening prior to surgery; muscle relaxants working at the neuromuscular junction used for intubation and/or anesthesia administration for the surgical procedure prior to CTM administration; and sedatives (i.e., midazolam) used as a co-induction agent for the surgical procedure prior to CTM administration
6. Patients taking warfarin, lithium, combination of ACE-inhibitors and furosemide
7. Patients with anemia (active clinically significant) and/or a history or evidence of asthma or heart failure
8. History of allergy or hypersensitivity to any component of Caldolor, aspirin (or aspirin related products), NSAIDs, or COX-2 inhibitors
9. Pregnant or nursing
10. History of severe head trauma that required current hospitalization, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurysm or CNS mass lesion
11. Weigh less than 30kg
12. Have a history of congenital bleeding diathesis (eg hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
13. Have GI bleeding that required medical intervention within the previous 6 weeks (unless definitive surgery has been performed)
14. Have a platelet count less than 30,000mm3 determined within the 28 days prior to surgery
15. Pre-existing dependence on narcotics or known tolerance to opioids
16. Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions and to return for the required assessments
17. Refusal to provide written authorization for use and disclosure of protected health information
18. Be on dialysis, have oliguria or calculated creatinine clearance of less than 60 mL/min (calculated using the Cockcroft and Gault formula) determined within the 28 days prior to surgery
19. Inability to achieve hemostasis or inability to close surgical incision, prior to Operating Room discharge
20. Operative procedure includes organ transplant
21. Pre or intra-operative procedure utilized for the prevention of pre- or post-operative pain (i.e. epidural or nerve blocks)
22. Be receiving full dose anticoagulation therapy or Activated Protein C within 6 hours before dosing (Prophylaxis with subcutaneous heparin is acceptable)
23. Have received another investigational drug within the past 30 days
24. Be otherwise unsuitable for the study in the opinion of the investigator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - Cooper Green Hospital / Jefferson Clinic, Birmingham, Alabama
  - Medical Center East / Alabama Clinical Therapeutics, Birmingham, Alabama
  - Springhill Hospital / Wilmax Clinical Research, Inc., Mobile, Alabama
  - Mobile Infirmary Medical Center / Wilmax Clinical Research, Inc., Mobile, Alabama
  - Jackson Hospital / Drug Research and Analysis Corporation, Montgomery, Alabama
  - Baptist Medical Center South / Drug Research and Analysis Corporation, Montgomery, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Valley OB/GYN, Colton, California
  - Research Support Personnel LLC, Wichita, Kansas
  - Chandler Medical Center; Ken Muse Research, Lexington, Kentucky
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - Health First Medical Group, Fort Worth, Texas
- Royal Adelaide Hospital, Adelaide, Australia

REFERENCES:
- [Derived] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the medical practices and/or clinics of the investigator/sub-investigators.
Pre-assignment Details: A total of 319 participants were randomized into two treatment groups. Randomized participants were additionally stratified by age and weight; three participants were randomized to incorrect stratification categories. All 319 participants received at least one dose of clinical trial material.
Groups:
- Placebo: The first dose of intravenous placebo will be administered at approximately the initiation of skin closure, prior to discharge to the recovery room. Seven subsequent doses of intravenous placebo will be administered every 6 hours. After receiving 8 doses of intravenous placebo, intravenous placebo will continue to be administered every 6 hours up to 5 days post surgery if pain medication is still required and intravenous access is present. All participants were able to receive morphine until approximately 45 minutes before the end of surgery. At that time on only fentanyl will be allow until the end of the surgery. Upon discharge from the operating room, participants will have access to morphine upon patient request or delivered by patient controlled analgesia.
- 800 mg Intravenous Ibuprofen: The first dose of intravenous ibuprofen will be administered at approximately the initiation of skin closure, prior to discharge to the recovery room. Seven subsequent doses of intravenous ibuprofen will be administered every 6 hours. After receiving 8 doses of intravenous ibuprofen, intravenous ibuprofen will continue to be administered every 6 hours up to 5 days post surgery if pain medication is still required and intravenous access is present. All participants were able to receive morphine until approximately 45 minutes before the end of surgery. At that time on only fentanyl will be allow until the end of the surgery. Upon discharge from the operating room, participants will have access to morphine upon patient request or delivered by patient controlled analgesia.
Period: Overall Study
Arm/Group | Placebo | 800 mg Intravenous Ibuprofen
Started | 153 | 166
Completed | 153 | 166
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 800 mg Intravenous Ibuprofen | Total
Number analyzed (Participants) | 153 | 166 | 319
Age, Customized [Number; unit: participants]
  Less than or equal to 45 years | 104 | 110 | 214
  45 to 70 years of age | 49 | 56 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 166 | 319
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 52 | 71 | 123
  Black or African American | 91 | 84 | 175
  Hispanic | 8 | 11 | 19
  Asian | 0 | 0 | 0
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 153 | 166 | 319
Weight [Number; unit: Kilograms]
  Less than or equal to 75 kilograms | 57 | 61 | 118
  Greater than 75 kilograms | 96 | 105 | 201

OUTCOME MEASURES:

1. Primary Outcome: Change in the Patient Demand for the Narcotic Analgesic, Morphine, Post Surgery
Description: Change in the amount of morphine use (in milligrams) by subjects in each treatment group for a 24 hour period post-surgery
Time Frame: 24 Hours
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Placebo | 800 mg Intravenous Ibuprofen
Number analyzed (Participants) | 153 | 166
milligrams | 57.0 (2.4) | 48.7 (2.3)

ADVERSE EVENTS:
Time Frame: 14 Days
Arm/Group | Placebo | 800 mg Intravenous Ibuprofen
Serious Adverse Events (participants affected / at risk) | 6/153 | 12/166
Other Adverse Events (participants affected / at risk) | 149/153 | 150/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | 800 mg Intravenous Ibuprofen (N=166)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peritoneal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Wound Dihisence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | 800 mg Intravenous Ibuprofen (N=166)
Nausea (Gastrointestinal disorders) | 85 (132) | 79 (137)
Flatulence (Gastrointestinal disorders) | 34 (41) | 42 (47)
Constipation (Gastrointestinal disorders) | 21 (21) | 13 (13)
Vomiting (Gastrointestinal disorders) | 12 (12) | 15 (18)
Pyrexia (General disorders) | 9 (9) | 6 (10)
Pruritis (Skin and subcutaneous tissue disorders) | 33 (51) | 32 (50)
Body temperature increased (Investigations) | 7 (10) | 7 (11)
Headache (Nervous system disorders) | 11 (14) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No